CLINICAL TRIAL: NCT02535910
Title: Fortification of Milk and Butter With Either vitaminD3 or 25(OH)D3: The Effect on Vitamin D Status and Cardiovascular Disease Risk Markers in Humans
Brief Title: Effect of vitaminD3 or 25(OH)D3 Fortified Dairy on Vitmain D Status and CVD Risk Markers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor Julie Lovegrove, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: VitD
Record Dates: First submitted 2015-07-28; First posted 2015-08-31 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Hypovitaminosis D; Cardiovascular Diseases
Keywords: vitamin D3; 25(OH)D3; vitamin D status; risk factors of cardiovascular diease
MeSH Terms: conditions — Vitamin D Deficiency; Cardiovascular Diseases | interventions — Cholecalciferol; Calcifediol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- breakfast rich in vitamin D3 (Experimental): subjects are asked to consume a breakfast with (20µg) vitamin D3 fortified milk and butter
  Interventions: Dietary Supplement: vitamin D3
- breakfast rich in 25(OH) D3 (Experimental): subjects are asked to consume a breakfast with (20µg) 25(OH) D3 fortified milk and butter
  Interventions: Dietary Supplement: 25(OH) D3
- Control (Placebo Comparator): subjects are asked to consume a normal milk and butter (no vitamin D is added) in the breakfast
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: vitamin D3 — Subjects are asked to consume a breakfast rich in 20 µg vitamin D3
  Other Names: cholecalciferol
  Arms: breakfast rich in vitamin D3
Dietary Supplement: 25(OH) D3 — Subjects are asked to consume a breakfast rich in 20 µg 25(OH)D3
  Other Names: calcifediol
  Arms: breakfast rich in 25(OH) D3
Dietary Supplement: Control — Subjects are asked to consume a breakfast without vitamin D
  Arms: Control

SUMMARY:
This study aims to compare the acute effect of consuming milk and butter fortified with either vitamin D3 or 25 (OH) D3 on serum/plasma vitamin D status in humans. In addition, the effect of vitamin D3 or 25 (OH) D3 in milk and butter on certain CVD risk markers and cognitive function will be examined.

DETAILED DESCRIPTION:
There is mounting evidence to show that vitamin D deficiency may increase the risk of many common and serious diseases, including osteoporosis, cardiovascular disease, some cancers and type 1 diabetes (Holick and Chen, 2008). Hypovitaminosis D is now prevalent in the UK general population. Due to diet and lifestyle changes and the use of sun block products most people do not endogenously synthesise sufficient vitamin D from sunlight exposure (Hyppönen and Power, 2007). Therefore, vitamin D intakes from dietary sources have become very important, however this is limited as there are only a few foods naturally rich in vitamin D.

Some countries (e.g. USA, Canada) fortify milk with vitamin D which results in milk being the major contributor to vitamin D intake. Vitamin D3 is the most common form used for the fortification of currently fortified foods. However, there is now some evidence that 25(OH)D3 can increase vitamin D status of humans more effectively than vitamin D3 (Bischoff-Ferrari et al, 2012; Cashman et al, 2012). To our knowledge, very few human intervention studies have compared the efficacy of 25(OH)D3 versus vitamin D3 to increase vitamin D status, and there has been no acute human study to examine the effect of the both forms of vitamin D fortified dairy products on vitamin D status in humans.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 20-35 kg/m2
* Glucose <7 mmol/l (not diagnosed with diabetes)
* Total cholesterol <7 mmol/l
* TAG <4 mmol/l
* Serum 25(OH)D3 ≤50 nmol/L
* Normal liver and kidney function
* Haemoglobin: adult male >125 g/L

Exclusion Criteria:

* Milk allergy/intolerance or lactose intolerance
* Cardiovascular, renal, gastrointestinal, respiratory, endocrine disease or cancer
* Use of nutritional supplements, particularly those containing vitamin D
* Outdoor workers and use of tanning beds
* Overseas holidays two months before or during study period

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the concentrations of vitamin D3, 25(OH)D3, 1, 25(OH)2D3 of the blood | Acute study: measured at 0 (baseline), 30, 60, 90, 120, 180, 240, 300, 360, 420, 480 min and 24 hour
Change from baseline in the concentrations of vitamin D3 and 25(OH)D3 of the chylomicron | Acute study: measured at 0 (baseline), 3, 6, 8 hour

SECONDARY OUTCOMES:
change from baseline in vascular reactivity measured by Endo-PAT | Acute study: measured at 0 (baseline) and the 24 hour
change from baseline in vascular reactivity measured by digital volume pulse (DVP) | Acute study: measured at 0 (baseline), 120, 240, 360, 480 min and 24 hour
change from baseline in plasma lipids (primarily triacylglycerol, apolipoprotein B, apolipoprotein B-48, apolipoprotien B-100, total-cholesterol, HDL-cholesterol, non-esterified fatty acids) | from 0 to 24 hour, but different measured time points for diferent lipids
  non-esterified fatty acids, apolipoprotein B, apolipoprotein B-48, apolipoprotein B-100 are taken at 0(baseline), 60, 120, 240, 360, 480 min and 24 hour; triacylglycerol is taken at 0, 30, 60, 90, 120, 180, 240, 300, 360, 420, 480 min and 24 hour; total and HDL-cholesterol only be measured at 0 (baseline)
change from baseline in markers of insulin resistance (glucose and insulin) | Acute study: measured at 0, 30, 60, 90, 120, 180, 240, 300, 360, 420, 480 min and 24 hour
change from baseline in nitric oxide | Acute study: measured at 0, 60, 120, 240, 360, 480 min and 24 hour
change from baseline in inflammatory markers (tumor necrosis factor alpha, C-reactive protein and interleukin 6) of the blood | Acute study: measured at 0, 60, 120, 240, 360, 480 min and 24 hour
change from baseline in blood pressure | Acute study: measured at 0, 120, 240, 360, 480 min and 24 hour
change from baseline in cognitive test | Acute study: measured at 0, 480 min and 24 hour
  Trail Making Test (TMT) will be used for cognitive test, which can provides information on visual search, scanning, speed of processing, mental flexibility, and executive function. The TMT consists of two parts: TMT-A requires a participant to draw lines sequentially connecting 25 encircled numbers distributed on a computer screen, whilst in the TMT-B the participant must alternate between numbers and letters (e.g., 1, A, 2, B, 3, C, etc.). TMT-A and TMT-B will be administered using a laptop computer. Results from this two tasks reported as the number of seconds required to complete the task (completion time). The longer time spent reveal greater cognitive impairment."

CONTACTS AND LOCATIONS:
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Guo J, Jackson KG, Che Taha CSB, Li Y, Givens DI, Lovegrove JA. A 25-Hydroxycholecalciferol-Fortified Dairy Drink Is More Effective at Raising a Marker of Postprandial Vitamin D Status than Cholecalciferol in Men with Suboptimal Vitamin D Status. J Nutr. 2017 Nov;147(11):2076-2082. doi: 10.3945/jn.117.254789. Epub 2017 Sep 20. PMID 28931588